CLINICAL TRIAL: NCT05156437
Title: Postoperative Antibiotic Management Duration Following Surgery for Intravenous Drug Abuse (IVDA) Endocarditis (OPTIMAL)
Acronym: OPTIMAL
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Vinay Badhwar (Other)
Responsible Party: Sponsor-Investigator, Vinay Badhwar, Executive Chair, Heart & Vascular Institute, West Virginia University
Organization: West Virginia University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2109416021
Record Dates: First submitted 2021-11-16; First posted 2021-12-14 (Actual); Last update posted 2023-12-07 (Actual); Status verified 2023-12

CONDITIONS: Endocarditis
Keywords: Intravenous Drug Abuse Endocarditis; Oral Antibiotics; IV Antibiotics
MeSH Terms: conditions — Endocarditis | interventions — Amoxicillin; Cephalexin; Dicloxacillin; Linezolid; Levofloxacin; Rifampin; Ampicillin; Oxacillin; Vancomycin; Daptomycin; Ceftriaxone; Cefepime; Ceftaroline

STUDY DESIGN:
Intervention Model Description: Postoperative patients who have undergone valvar repair or replacement for IVDA endocarditis will be randomized into two arms: Experimental: 2 weeks of postoperative inpatient IV antibiotic therapy followed by 4 weeks of oral therapy with outpatient follow-up; Control: conventional 2 weeks of postoperative inpatient IV antibiotic therapy followed by 4 weeks of IV antibiotic therapy (inpatient or facility supervised if indwelling catheter utilized).
  Both groups will receive aggressive drug rehabilitation with mandatory participation in a formal psychiatric rehabilitation program for a minimum of 6 weeks (combined inpatient and outpatient), will be followed by Infectious Disease, will undergo monitoring of treatment efficacy with serum antibiotic levels, will undergo surveillance monitoring of treatment efficacy with blood cultures, will participate in a compliance tracking tool for medication administration (e.g. a centrally managed core site mobile Medisafe compliance program.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group I (Experimental) (Experimental): Two (2) weeks of postoperative inpatient IV antibiotic therapy followed by four (4) weeks of oral therapy with outpatient follow-up.
  Interventions: Drug: Amoxycillin, Cefalexin, Dicloxacillin, Linezolid, Levofloxacin, Rifampicin; Drug: Ampicillin, Oxacillin, Vancomycin, Daptomycin, Ceftriaxone, Cefepime, Ceftaroline
- Group II (Control Group) (Active Comparator): Conventional two (2) weeks of postoperative inpatient IV antibiotic therapy followed by four (4) weeks of IV antibiotic therapy (inpatient or facility supervised if indwelling catheter utilized).
  Interventions: Drug: Ampicillin, Oxacillin, Vancomycin, Daptomycin, Ceftriaxone, Cefepime, Ceftaroline

INTERVENTIONS:
Drug: Amoxycillin, Cefalexin, Dicloxacillin, Linezolid, Levofloxacin, Rifampicin — Amoxycillin, Cefalexin, Dicloxacillin, Linezolid, Levofloxacin, Rifampicin
  Arms: Group I (Experimental)
Drug: Ampicillin, Oxacillin, Vancomycin, Daptomycin, Ceftriaxone, Cefepime, Ceftaroline — Ampicillin, Oxacillin, Vancomycin, Daptomycin, Ceftriaxone, Cefepime, Ceftaroline

SUMMARY:
The purpose of this study is to determine the safety and compliance of initial intravenous (IV) antibiotics followed by oral antibiotic therapy following uncomplicated IVDA endocarditis. Endocarditis has a high rate of sickness and death, involves a long hospitalization and a long-term use of IV antibiotics necessitating six (6) weeks of in-patient hospital stay, and comes with a high cost.

ELIGIBILITY:
Inclusion Criteria:

* The age of the patient is ≥ 18.
* The patient has undergone an urgent or emergent primary cardiac valvar operation as treatment for IVDA endocarditis, with blood cultures positive for Streptococcus, Enterococcus faecalis, Staphylococcus aureus, or coagulase-negative Staphylococci
* The patient has received 2 weeks of postoperative inpatient IV antibiotic therapy with negative blood cultures and no residual active infection by imaging (i.e. computerized axial tomography, echocardiography)
* The patient has the capacity to participate in a compliance tracking tool for medication administration (e.g. a centrally managed core site mobile Medisafe compliance https://www.medisafe.com/) as confirmed by both a physician and a care management team member

Exclusion Criteria:

* Inability to give informed consent
* Residual infection requiring IV antibiotic therapy
* Any persistent secondary noncardiac infection (e.g. infections of solid organs or joints)
* Known poor compliance or deemed incapable to comply with the compliance tracking tool
* Reduced absorption or inability to receive oral treatment due to a gastrointestinal disorder
* Any infection involving a more virulent organisms, such as fungal infections or infections with Serratia or HACEK infections (Haemophilus, Aggregatibacter, Cardiobacterium, Eikenella, Kingella).
* Cancer not otherwise in remission or in need of current or future oncologic therapy
* Medically immunocompromised state
* Reoperative valvar operation for IVDA endocarditis
* History of habitual noncompliance
* Pregnancy
* Mental incapacity
* Unable to perform local or institutional medical and psychiatric follow up
* Unstable home environment
* Inadequate access to mobile cell service (geographic/rurality)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-03-16 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
To assess all-cause mortality at six (6) months post-surgery. | Six months
  To assess all-cause mortality at six (6) months post-surgery.
To assess all-cause mortality at (12) months post-surgery. | One year
  To assess all-cause mortality at (12) months post-surgery.
To assess recurrent blood culture positive infection. | Six months
  To assess recurrent blood culture positive infection.
To assess recurrent blood culture positive infection. | One year
  To assess recurrent blood culture positive infection.
To assess cardiac re-operation. | Six months
  To assess cardiac re-operation.
To assess cardiac re-operation. | One year
  To assess cardiac re-operation.

SECONDARY OUTCOMES:
Readmission for recurrent infection or cardiac re-operation | Six months
  Readmission for recurrent infection or cardiac re-operation
Readmission for recurrent infection or cardiac re-operation | One year
  Readmission for recurrent infection or cardiac re-operation
Cost of care | Through study completion, an average of one year
  Cost of care

CONTACTS AND LOCATIONS:
Overall Officials: Vinay Badhwar, MD, Principal Investigator — West Virginia University
Locations (1):
- WVU Heart and Vascular Institute, Morgantown, West Virginia, United States

REFERENCES:
- [Background] Iversen K, Ihlemann N, Gill SU, Madsen T, Elming H, Jensen KT, Bruun NE, Hofsten DE, Fursted K, Christensen JJ, Schultz M, Klein CF, Fosboll EL, Rosenvinge F, Schonheyder HC, Kober L, Torp-Pedersen C, Helweg-Larsen J, Tonder N, Moser C, Bundgaard H. Partial Oral versus Intravenous Antibiotic Treatment of Endocarditis. N Engl J Med. 2019 Jan 31;380(5):415-424. doi: 10.1056/NEJMoa1808312. Epub 2018 Aug 28. PMID 30152252
- [Background] Spellberg B, Chambers HF, Musher DM, Walsh TL, Bayer AS. Evaluation of a Paradigm Shift From Intravenous Antibiotics to Oral Step-Down Therapy for the Treatment of Infective Endocarditis: A Narrative Review. JAMA Intern Med. 2020 May 1;180(5):769-777. doi: 10.1001/jamainternmed.2020.0555. PMID 32227127
- [Background] Lemaignen A, Bernard L, Tattevin P, Bru JP, Duval X, Hoen B, Brunet-Houdard S, Mainardi JL, Caille A; RODEO (Relais Oral Dans le traitement des Endocardites a staphylocoques ou streptOcoques) and AEPEI (Association pour l'Etude et la Prevention de l'Endocardite Infectieuse) study groups. Oral switch versus standard intravenous antibiotic therapy in left-sided endocarditis due to susceptible staphylococci, streptococci or enterococci (RODEO): a protocol for two open-label randomised controlled trials. BMJ Open. 2020 Jul 14;10(7):e033540. doi: 10.1136/bmjopen-2019-033540. PMID 32665381
- [Background] Brown E, Gould FK. Oral antibiotics for infective endocarditis: a clinical review. J Antimicrob Chemother. 2020 Aug 1;75(8):2021-2027. doi: 10.1093/jac/dkaa106. PMID 32240296
- [Background] Scholl L, Seth P, Kariisa M, Wilson N, Baldwin G. Drug and Opioid-Involved Overdose Deaths - United States, 2013-2017. MMWR Morb Mortal Wkly Rep. 2018 Jan 4;67(5152):1419-1427. doi: 10.15585/mmwr.mm675152e1. PMID 30605448
- [Background] Wurcel AG, Anderson JE, Chui KK, Skinner S, Knox TA, Snydman DR, Stopka TJ. Increasing Infectious Endocarditis Admissions Among Young People Who Inject Drugs. Open Forum Infect Dis. 2016 Jul 26;3(3):ofw157. doi: 10.1093/ofid/ofw157. eCollection 2016 Sep. PMID 27800528
- [Background] Kornbau C, Lee KC, Hughes GD, Firstenberg MS. Central line complications. Int J Crit Illn Inj Sci. 2015 Jul-Sep;5(3):170-8. doi: 10.4103/2229-5151.164940. PMID 26557487
- [Background] Badhwar V, Wei LM, Rankin JS. Seeing the entire forest in endocarditis. J Thorac Cardiovasc Surg. 2016 Sep;152(3):681-2. doi: 10.1016/j.jtcvs.2016.05.050. Epub 2016 Jun 4. No abstract available. PMID 27325495
- See also: Centers for Disease Control and Prevention Wide-ranging Online Data for Epidemiologic Research (CDC WONDER): Multiple cause of death 1999-2017 — http://wonder.cdc.gov